CLINICAL TRIAL: NCT06106789
Title: A Study of the Clinical Benefit of Tobramycin Inhalation Solution
Status: Active, not recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Rui Yang, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYX-YR-20230101
Record Dates: First submitted 2023-10-16; First posted 2023-10-30 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Bronchiectasis; Cystic Fibrosis; Lung Infection
Keywords: Bronchiectasis; Cystic Fibrosis; Lung Infection; Tobramycin inhalation solution; Antimicrobial non-nebulized inhalation preparations; Safety; Efficacy; Economical
MeSH Terms: conditions — Bronchiectasis; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Bronchiectasis: 1. Patients with a past medical history or a diagnosis of bronchiectasis in the current case;
  2. Patients seen or admitted to the hospital from 1 January 2021 to 31 December 2023 (including outpatient, emergency, and inpatient);
  3. Case record of at least 1 course of treatment (continuous administration for 28 days) with tobramycin inhalation solution or other antibiotic nebulisation;
  4. Patients with a positive copper-green test at the first visit.
  Interventions: Drug: Tobramycin inhalation solution
- Cystic fibrosis: 1. Patients with a past medical history or a diagnosis of cystic fibrosis in the current case;
  2. Patients who were seen or admitted to the hospital from 1 January 2021 to 31 December 2023 (including outpatient, emergency, and inpatient);
  3. Case record of at least 1 course of treatment (continuous administration for 28 days) with tobramycin inhalation solution or other antibiotic nebulisation;
  4. Patients with a positive copper-green test at the first visit.
  Interventions: Drug: Tobramycin inhalation solution
- Multidrug-resistant bacterial lung infections: 1. Patients with a diagnosis of pulmonary infection;
  2. Patients admitted to the hospital from 1 January 2021 to 31 December 2023 (only inpatients were included);
  3. Case records with completion of at least 3 days of treatment with tobramycin inhalation solution or other antibiotic nebulisation;
  4. The patient tested positive for pathogens at least once during the period of medication.
  Interventions: Drug: Tobramycin inhalation solution

INTERVENTIONS:
Drug: Tobramycin inhalation solution — Tobramycin Inhalation Solution is a yellowish clear liquid, the main ingredient is tobramycin.
  Antimicrobial non-nebulized inhalation preparation according to the current clinical situation, mainly polymyxin, amikacin, depending on the specific circumstances of each hospital.
  Other Names: Antimicrobial non-nebulized inhalation preparations

SUMMARY:
This project will use literature analysis, expert research, real-world data mining and other methods to investigate the current status of the application of antimicrobial aerosolized inhalation in healthcare institutions, combine expert recommendations and real-world data analysis results to explore potential risk points in the process of antimicrobial aerosolized drug delivery, and sort out the key points of drug use management in healthcare institutions and the key points of regulatory recommendations for healthcare institutions.

DETAILED DESCRIPTION:
The current status of nebulised inhalation of antimicrobial drugs was examined by the main subject through literature search and expert research. The researchers selected patients who visited or were admitted to Qianfoshan Hospital in Shandong Province during the period from 1 January 2021 to 31 December 2023, extracted data according to the inclusion and exclusion criteria, and used tobramycin inhalation solution as the study group, and injectable antimicrobials used by inhalation such as amikacin, polymyxin E sodium methanesulfonate, polymyxin E sulphate, polymyxin B sulphate and other antimicrobials in a multicentre real-world cohort study as the control group, and adopted a multi A multi-centre real-world cohort study was conducted to examine the effectiveness, safety and economy of nebulised inhalation of antimicrobial drugs in different levels of healthcare institutions in China, to directly compare the risk of use of injectable over-the-counter nebulised inhalation with that of inhalation formulations, and also to provide post-marketing re-evaluation for the newly marketed tobramycin inhalation solution and to provide evidence-based evidence for the rational use of medication in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis

  1. Patients with a past medical history or a diagnosis of bronchiectasis in the current case;
  2. Patients seen or admitted to the hospital from 1 January 2021 to 31 December 2023 (including outpatient, emergency, and inpatient);
  3. Case record of at least 1 course of treatment (continuous administration for 28 days) with tobramycin inhalation solution or other antibiotic nebulisation;
  4. Patients with a positive copper-green test at the first visit.
* Cystic fibrosis

  1. Patients with a past medical history or a diagnosis of cystic fibrosis in the current case;
  2. Patients who were seen or admitted to the hospital from 1 January 2021 to 31 December 2023 (including outpatient, emergency, and inpatient);
  3. Case record of at least 1 course of treatment (continuous administration for 28 days) with tobramycin inhalation solution or other antibiotic nebulisation;
  4. Patients with a positive copper-green test at the first visit.
* Multidrug-resistant bacterial lung infections

  1. Patients with a diagnosis of pulmonary infection;
  2. Patients admitted to the hospital from 1 January 2021 to 31 December 2023 (only inpatients were included);
  3. Case records with completion of at least 3 days of treatment with tobramycin inhalation solution or other antibiotic nebulisation;
  4. The patient tested positive for pathogens at least once during the period of medication.

Exclusion Criteria:

* Bronchiectasis Patients with key information missing from the study, such as therapeutic agents, diagnostic information for bronchiectasis, etc.
* Cystic fibrosis Patients with cystic fibrosis, for which key information is missing, such as treatment medication, diagnosis of cystic fibrosis.
* Multidrug-resistant bacterial lung infections Patients hospitalized with severe pneumonia were missing key study information, such as laboratory tests not performed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen or admitted to the hospital (including outpatient, emergency, and inpatient) from January 1, 2021 - December 31, 2023, including:
  1. Patients with bronchiectasis combined with P. aeruginosa infection: nebulized inhaled antimicrobials to clear pathogens or to reduce pathogen load;
  2. Patients with cystic fibrosis combined with P. aeruginosa infection: nebulized inhaled antimicrobials to clear pathogens or to reduce pathogen load;
  3. Patients with multidrug-resistant bacterial lung infections using inhaled antimicrobials as an adjunctive therapeutic regimen to intravenous administration.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Total Adverse Reaction Incidence Rate | Through study completion，up to half a year.
  To evaluate the safety of injectable over-the-counter nebulized inhalation versus inhalation formulations by analyzing the incidence of total adverse reactions, and to provide first-line, real-world data to support post-market re-evaluation.
Pathogen clearance | Through study completion，up to half a year.
  To evaluate the effectiveness of the clinical application of injectable over-the-counter nebulized inhalation versus inhalation formulations by analyzing the pathogen clearance rate, and to provide first-line real-world data support for post-market re-evaluation of the product.
Average hospitalization cost per visit | Through study completion，up to half a year.
  To provide first-line, real-world data support for post-market re-evaluation of the product by analyzing the average per-hospitalization cost to evaluate the economics of the clinical application of injectable over-the-counter nebulized inhalation versus inhalation formulations.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Yang, MD, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Rui Yang,MD, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No